CLINICAL TRIAL: NCT02609581
Title: Non-Interventional Study (NIS) on the Tolerability of Sublingual Immunotherapy With LAIS® Mites Tablets in Consideration of the Chosen Titration Schedule in Everyday Practice
Brief Title: Tolerability of SLIT With LAIS® Mites Allergoid Tablets
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ralph Mösges, Prof. Dr. Ralph Mösges, University Hospital of Cologne
Other Study IDs: LF HDM/Titra/2015/D
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Allergic Rhinitis
Keywords: Non Interventional Study; NIS; sublingual immunotherapy; allergen; Mites
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy; Tablets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sublingual Immunotherapy with tablets (mites) — Sublingual immunotherapy involves putting a tablet of allergen extracts (mites) under the tongue to swallow the extract.
  Other Names: Sublingual immunotherapy

SUMMARY:
To expand knowledge on the application and tolerability of immunotherapy with LAIS® Mites allergoid tablets as well as knowledge on the alleviation of symptoms during sublingual therapy in special consideration of the chosen titration schedule in everyday practice.

DETAILED DESCRIPTION:
Until now, results from controlled studies with their specific requirements (patient selection, defined inclusion and exclusion criteria, close patient management and monitoring, randomisation) are available for LAIS® Mites allergoid tablets only for a small patient population. In addition, an open-label, controlled study and an observational study have been carried out investigating the clinical efficacy and tolerability of the preparation. Owing to the differences in the study designs, the allergen dose administered and the frequency with which the preparation was applied varied among the individual studies, making it necessary to gather further data on the safety and tolerability of the preparation in a larger patient population.

The observation schedule of this NIS (NIS in accordance with Article 67 Paragraph 6 of the German Medicinal Products Act (AMG)), which takes into account the recommendations made by the German Federal Institute for Drugs and Medical Devices (BfArM) and by the Paul Ehrlich Institute for planning, implementing and evaluating an NIS, is geared to the routine procedure carried out for patients with allergies to tree pollen.

The aim of this observational study is to observe and document the tolerability and improvement of symptoms after treatment with LAIS® Mites allergoid tablets under normal application conditions and in consideration of the chosen titration schedule in therapeutic practice - in accordance with the patient information leaflet - in a large patient population:

Retrospective survey of rhinitis/rhinoconjunctivitis symptoms induced by tree pollen Overall symptomatology Documentation of restrictions caused by allergy/asthma Tolerability of the treatment by means of AE documentation Patient compliance

Additional requirements extending beyond the specifications listed in the patient information leaflet on product use, patient groups, dosage, contraindications, etc., will not be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older having allergies within the scope of specifications stated in the patient information leaflet

Exclusion Criteria:

* Contraindications according to the patient information leaflet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older can be enrolled in the NIS if sublingual specific immunotherapy has been indicated due to allergic rhinoconjunctivitis or allergic bronchial asthma induced by the allergens to be investigated (mites).
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment of the tolerability of SLIT with LAIS® mites allergoid tablets on the description of adverse events and serious adverse events. | 13 month
  The description of adverse events/serious adverse events (AE/SAE) encompasses frequency, intensity, duration, relationship to LAIS® mites tablets and actions taken due to the treatment with LAIS® mites tablets and other concomitant medication. The documentation of adverse events takes place at visit 1, at visit 2 (after titrationphase) and at visit 3 (after first year of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Prof. Dr., Principal Investigator — University Hospital Cologne

IPD SHARING:
Plan to Share IPD: No